CLINICAL TRIAL: NCT05288556
Title: Single Site, Prospective, Phase I Study, Safety and Efficacy of Enteral Feeding Tube Stoma Site Accessory
Brief Title: Safety and Efficacy of Enteral Feeding Tube Stoma Site Accessory
Acronym: SSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Voluntary pause in enrollment to revise inclusion criteria and need for reliable transportation, after one unanticipated problem with a participant who had challenges attending safety clinical visits.
Sponsor: Eric Yudelevich (Other)
Responsible Party: Sponsor-Investigator, Eric Yudelevich, Eric Yudelevich, MD Assistant Professor, Director of Clinical Competency Development, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-143
Record Dates: First submitted 2022-02-03; First posted 2022-03-21 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Feeding Tube Complication

STUDY DESIGN:
Intervention Model Description: Single Site, Prospective, Phase I Study, Safety and Efficacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stoma Site Accessory (Experimental): Stoma site accessory with enteral tube replacement procedure.
  Interventions: Device: Placement of stoma site enteral feeding tube accessory

INTERVENTIONS:
Device: Placement of stoma site enteral feeding tube accessory — The study stoma site accessory will be attached at the stoma site during an enteral tube replacement procedure the patient is scheduled to have as a standard of care procedure. The study stoma site accessory is compatible with commercially available enteral nutrition feeding tubes ranging from size 16 to 20 French tubing that are adjustable to variable length.

SUMMARY:
The purpose of the study is to collect safety and efficacy data on the performance of the study stoma site accessory when used to prevent abdominal wall leakage for patients with a long term feeding tube.

This accessory has been developed by the Cleveland Clinic and will be used for the first time in human subjects according to the labeled indication for clinical use in accordance with the Manufacturer's Instructions for Use based on other similar, FDA approved gastrostomy and jejunostomy enteral feeding tube accessory components.

After providing informed consent, eligible patients will receive a study stoma site accessory during a feeding tube replacement procedure the patient is scheduled to have as a standard of care procedure.

DETAILED DESCRIPTION:
The purpose of the study is to collect safety and efficacy data on the performance of the study stoma site accessory when used to prevent abdominal wall leakage for patients with a long term, ≥ 3 months, enteral feeding tube including, gastrostomy or jejunostomy tubes. This study accessory has been developed by the Cleveland Clinic (CC) for clinical use in human subjects and will be used according to the labeled indication and in accordance with the Manufacturer's Instructions for Use based on other similar, Food and Drug Administration (FDA) approved enteral tube stoma site accessory components. Patients receiving the study accessory will also be asked pre-procedure and post-procedure quality of life questions to identify change in quality of life. After providing informed consent, eligible patients will receive a study stoma site accessory during an upcoming enteral tube replacement procedure the patient is scheduled to have as a standard of care procedure.

The study stoma site accessory, for regulatory purposes, can be considered an accessory to a newly replaced feeding tube. The accessory materials and method of use are substantially similar to commercially available feeding tubes used with percutaneous endoscopic gastrostomy (PEG), percutaneous endoscopic gastrojejunostomy (PEGJ) and direct percutaneous endoscopic jejunostomy (DPEJ). We believe that, since the study stoma site accessory attaches to the external portion of a newly replaced feeding tube at a previously established stoma site and inserts 1 cm into the stoma, which is not as deep as the actual feeding tube, it poses no significant risk to its users. By potentially decreasing the leakage from the edges of the tube and the friction of the tube against the skin, it does not pose a risk of local infection. It is made of commercially available, FDA cleared materials commonly used for enteral feeding tubes and tube components that the patient already has in place. The study accessory will be sterilized and packaged at the Cleveland Clinic through a validated process and provided specific numerical identification for documented tracking.

This study will evaluate the safety and efficacy of the study stoma site accessory used in place of a commercially available feeding tube accessory, i.e., button or flange, at the time of a standard of care replacement procedure the patient is scheduled to have at Cleveland Clinic's Main Campus. Patients enrolled in the study will participate for a period of 6 months with outcomes assessed using our protocol patient questionnaires. The length of the study will be approximately 12-18 months to allow for recruitment, and 6 months of ongoing follow-up after the last patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged ≥22 and ≤85 Note: Because the study accessory is designed for adult use participants <22 years of age are excluded but will be eligible for future trials, if applicable
* Ability to understand and the willingness to sign a written informed consent document
* Patients with existing gastrostomy and jejunostomy enteral feeding tubes, placed ≥ 3 months, undergoing replacement of feeding tube inpatient or outpatient
* Willing to adhere to placement of study stoma site accessory and ability to take oral temperature at specified times
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Willing to adhere to removal of study stoma site accessory at month 6

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patient requires general anesthesia in an OR for tube changes
* Current use of steroids (any dose) daily ≥ 3 months including, but not limited to: prednisone, prednisolone, methylprednisolone, cyclosporine
* Current use of Immunosuppressants including, but not limited to: azathioprine, mycophenolate.
* BMI ≥ 40
* Non-English speaking patients
* Pregnant Women
* Known allergic reactions to components of the study stoma site accessory [Medical Grade Silicone]
* Treatment with another investigational drug or device within 6 months of screening/baseline
* Uncontrolled illness, recent open abdominal surgery or social situations that in the opinion of the investigative team would limit compliance with study requirements, including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness
  * Unable to self-report
  * Not ambulatory and incapable of carrying out all self-care
  * Unsuccessful stoma site study accessory placement at time of initial replacement procedure

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yudelevich, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeLegge RL, DeLegge MH. Percutaneous endoscopic gastrostomy evaluation of device materials: are we "failsafe"? Nutr Clin Pract. 2005 Dec;20(6):613-7. doi: 10.1177/0115426505020006613. PMID 16306298
- [Background] ASGE Technology Committee; Kwon RS, Banerjee S, Desilets D, Diehl DL, Farraye FA, Kaul V, Mamula P, Pedrosa MC, Rodriguez SA, Varadarajulu S, Song LM, Tierney WM. Enteral nutrition access devices. Gastrointest Endosc. 2010 Aug;72(2):236-48. doi: 10.1016/j.gie.2010.02.008. Epub 2010 Jun 11. PMID 20541746
- [Background] Green SM, Townsend K, Jarrett N, Fader M. The experiences and support needs of people living at home with an enteral tube: a qualitative interview study. J Hum Nutr Diet. 2019 Oct;32(5):646-658. doi: 10.1111/jhn.12656. Epub 2019 Apr 21. PMID 31006929
- [Background] Malik F, Baig SN, Patel B, Gonzalez M, Nfonoyim J. Unusual complication of a percutaneous gastrostomy tube. J Community Hosp Intern Med Perspect. 2019 Sep 5;9(4):325-326. doi: 10.1080/20009666.2019.1650410. eCollection 2019. PMID 31528280
- [Background] Potack JZ, Chokhavatia S. Complications of and controversies associated with percutaneous endoscopic gastrostomy: report of a case and literature review. Medscape J Med. 2008 Jun 17;10(6):142. PMID 18679534
- [Background] Blumenstein I, Shastri YM, Stein J. Gastroenteric tube feeding: techniques, problems and solutions. World J Gastroenterol. 2014 Jul 14;20(26):8505-24. doi: 10.3748/wjg.v20.i26.8505. PMID 25024606
- [Background] Gramlich L, Hurt RT, Jin J, Mundi MS. Home Enteral Nutrition: Towards a Standard of Care. Nutrients. 2018 Aug 4;10(8):1020. doi: 10.3390/nu10081020. PMID 30081546
- [Background] Mundi MS, Pattinson A, McMahon MT, Davidson J, Hurt RT. Prevalence of Home Parenteral and Enteral Nutrition in the United States. Nutr Clin Pract. 2017 Dec;32(6):799-805. doi: 10.1177/0884533617718472. Epub 2017 Jul 17. PMID 28715295
- [Background] Ojo O, Keaveney E, Wang XH, Feng P. The Effect of Enteral Tube Feeding on Patients' Health-Related Quality of Life: A Systematic Review. Nutrients. 2019 May 10;11(5):1046. doi: 10.3390/nu11051046. PMID 31083338
- [Background] Hall BT, Englehart MS, Blaseg K, Wessel K, Stawicki SP, Evans DC. Implementation of a dietitian-led enteral nutrition support clinic results in quality improvement, reduced readmissions, and cost savings. Nutr Clin Pract. 2014 Oct;29(5):649-55. doi: 10.1177/0884533614538285. PMID 25606646

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential patients were recruited based on physician referrals at 2 of Cleveland Clinic's academic medical centers between 4/29/22 and 6/22/23.
  Of the 31 patients screened for eligibility, five patients were consented and scheduled for the study stoma accessory during a standard of care replacement procedure. Of these five, one retained the accessory into week six and two retained the accessory up to week 12 of the 24 week study period.
Period: Overall Study
Arm/Group | Stoma Site Accessory
Started | 5
Completed | 3 (Patients were asked to complete pre procedure patient reported outcomes and to take their oral temperature daily for the first ten days. They were scheduled for the week two post procedure research follow up visit to assess safety and efficacy of the stoma accessory.)
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Successful Accessory Placement
Description: Using the accessory placement date as the baseline, the number of participants with study accessory still in place will be measured at week 2.
  The measurement tool is a question the patients will be asked to determine "Is the device still in place?" The response is captured in a database with the answers "Yes" or "No."
Time Frame: Week 2 Visit
Population: Four of five participants successfully completed the stoma accessory placement procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Successful Accessory Placement
Description: Using the accessory placement date as the baseline, the number of participants with study accessory still in place will be measured at week 4.
  The measurement tool is a question the patients will be asked to determine "Is the device still in place?" The response is captured in a database with the answers "Yes" or "No."
Time Frame: Week 4 Phone call
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 4
Participants | 3

3. Primary Outcome: Successful Accessory Placement
Description: Using the accessory placement date as the baseline, the number of participants with study accessory still in place will be measured at week 6.
  The measurement tool is a question the patients will be asked to determine "Is the device still in place?" The response is captured in a database with the answers "Yes" or "No."
Time Frame: Week 6 Phone call
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 4
Participants | 3

4. Primary Outcome: Successful Accessory Placement
Description: Using the accessory placement date as the baseline, the number of participants with study accessory still in place will be measured at month 3.
  The measurement tool is a question the patients will be asked to determine "Is the device still in place?" The response is captured in a database with the answers "Yes" or "No."
Time Frame: Month 3 Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 4
Participants | 2

5. Primary Outcome: Successful Accessory Placement
Description: Using the accessory placement date as the baseline, the number of participants with study accessory still in place will be measured at month 4.
  The measurement tool is a question the patients will be asked to determine "Is the device still in place?" The response is captured in a database with the answers "Yes" or "No."
Time Frame: Month 4 Visit
Population: No participant reached the 4 month mark, as described previously (and captured under Early Termination).
  Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

6. Primary Outcome: Successful Accessory Placement
Description: Using the accessory placement date as the baseline, the number of participants with study accessory still in place will be measured at month 6.
  The measurement tool is a question the patients will be asked to determine "Is the device still in place?" The response is captured in a database with the answers "Yes" or "No."
Time Frame: Month 6 Visit
Population: No participant reached the 6 month time point as described previously (and captured under Early Termination). Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

7. Primary Outcome: Number of Participants With a Feeding Tube Complication With a Study Accessory
Description: Minor complications associated with feeding tubes as defined by clinical assessment of treating physician at week baseline. Total number of complications will be reported per patient at each time point.
Time Frame: Baseline
Population: No complications at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 5
Participants | 0

8. Primary Outcome: Number of Participants With a Feeding Tube Complication With a Study Accessory
Description: Minor complications associated with feeding tubes as defined by clinical assessment of treating physician at week 2. Total number of new complications will be reported per patient at each time point.
Time Frame: Week 2 Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 5
Participants | 2

9. Primary Outcome: Number of Participants With a Feeding Tube Complication With a Study Accessory
Description: Minor complications associated with feeding tubes as defined by clinical assessment of treating physician at month 3. Total number of new complications will be reported per patient at each time point.
Time Frame: Month 3 Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 5
Participants | 1

10. Primary Outcome: Number of Participants With a Feeding Tube Complication With a Study Accessory
Description: Minor complications associated with feeding tubes as defined by clinical assessment of treating physician at early termination. Total number of new complications will be reported per patient at each time point.
Time Frame: Early termination (during the first 6 months)
Population: as for outcome 6
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

11. Primary Outcome: Number of Participants With a Feeding Tube Complication With a Study Accessory
Description: Minor complications associated with feeding tubes as defined by clinical assessment of treating physician at month 6. Total number of new complications will be reported per patient at each time point.
Time Frame: Month 6 Visit
Population: as for outcome 6
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

12. Secondary Outcome: Quality of Life Patient-Reported Outcomes Measurement Information System (PROMIS) 10 Questionnaire
Description: Using the PROMIS 10 questionnaire we will measure change using the physical and mental health global T scores for patient quality of life after intervention as self-reported by participants. Physical T score ranges 16.2 as the lowest to 67.7 as the highest and mental T score ranges from 21.2 to 67.6. A higher score at month 6 is indication of improvement.
Time Frame: Baseline
Population: Four of five participants completed the baseline PROMIS10 survey
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 4
T Score
  Mental Health | 45.125 (6.774646362)
  Physical Health | 44.075 (5.999097154)

13. Secondary Outcome: Quality of Life PROMIS 10 Questionnaire
Description: Using the PROMIS 10 questionnaire we will measure change using the global physical and global mental health T scores for patient quality of life after intervention as self-reported by participants. Physical T score ranges 16.2 as the lowest to 67.7 as the highest and mental T score ranges from 21.2 to 67.6. A higher score at termination is indication of improvement.
Time Frame: Early termination (during the first 6 months)
Population: Participants were asked to complete the PROMIS 10 at early termination whenever it occurred prior to month 6.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 3
T Score
  Physical Health | 45.6 (3.00499584)
  Mental Health | 43.5 (4.582575695)

14. Secondary Outcome: Quality of Life PROMIS 10 Questionnaire
Description: Using the PROMIS 10 questionnaire we will measure change using the global physical and global mental health T scores for patient quality of life at the 6 month time point, as self-reported by participants. No specific threshold is used. Physical T score ranges 16.2 as the lowest to 67.7 as the highest and mental T score ranges from 21.2 to 67.6. A higher score at month 6 is indication of improvement.
  No participant reached the 6 month mark, as described previously (and captured under Early Termination). Therefore, there are 0 PROMIS 10 scores to report.
  Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Time Frame: Month 6 Visit
Population: No patient reached the 6 month time point. No participant reached the 6 month time point as described previously (and captured under Early Termination). Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

15. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at baseline.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
Time Frame: Baseline
Population: Four of five participants completed this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 4
score on a scale | 10.25 (2.5)

16. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at week 2.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
Time Frame: Week 2 Visit
Population: Three of four participants completed this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 3
score on a scale | 12.33333333 (4.618802154)

17. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at week 4.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
Time Frame: Week 4 Phone Call
Population: Three of five patients completed this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 3
score on a scale | 16 (4.041451884)

18. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at week 6.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
Time Frame: Week 6 Phone Call
Population: Three of five participants completed this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 3
score on a scale | 11.66666667 (5.131601439)

19. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at month 3.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
Time Frame: Month 3 Visit
Population: Two of five participants completed this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 2
score on a scale | 16 (1.414213562)

20. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at early termination.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
Time Frame: Early Termination (during the first 6 months)
Population: Participants were asked to complete the Characteristics of Pain and Leakage at early termination whenever it occurred prior to month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 3
score on a scale | 14.66666667 (0.577350269)

21. Secondary Outcome: Characteristics of Pain and Leakage Questionnaire
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at month 4.
  Each question will have a score from one to 5 and the scores will be summed to a total score (with a total score of 4 representing lowest quality of life, and a score of 20 representing the highest quality of life)
  No participant reached the 4 month mark, as described previously (and captured under Early Termination). Therefore, there are 0 Characteristics of Pain and Leakage Questionnaire scores to report.
  Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Time Frame: Month 4 Visit
Population: No participant reached the 4 month mark, as described previously (and captured under Early Termination). Therefore, there are 0 Characteristics of Pain and Leakage Questionnaire scores to report.
  Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

22. Secondary Outcome: Characteristics of Pain and Leakage
Description: Using a novel Characteristics of Pain and Leakage questionnaire with 4 unique quality of life questions, investigators will collect patient self reported data at month 6.
  Each question will have a score from one to 5 and the scores will be summed to a total score. A higher score corresponds to a higher quality of life.
  No participant reached the 6 month mark, as described previously (and captured under Early Termination). Therefore, there are 0 Characteristics of Pain and Leakage Questionnaire scores to report. Please see the completed questionnaires captured by Early Termination on Outcome Measure #20.
  Outcome Measures is reported with zero total participants analyzed, because the study was terminated and data collection stopped prior to the pre-specified time points/end points for an outcome.
Time Frame: Month 6 Visit
Population: No participants completed month 6 outcomes measures.
Arm/Group | Stoma Site Accessory
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: If the Principal Investigator, or his/her designee concludes the study accessory is malfunctioning, inadvertently removed or compromised or, for any reason, determined to be a greater risk than benefit, e.g., the patient has an allergic reaction, and is replaced by a commercially available accessory, the patient will be exited from the study by early termination.
Arm/Group | Stoma Site Accessory
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stoma Site Accessory (N=5)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) — Patient admitted to be treated for infection in blood stream on date of elective surgical procedure unrelated to study.
Hospitalization (General disorders) | 1 (1) — Patient with history of vertigo and dizziness admitted through ED after falling, not related to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stoma Site Accessory (N=5)
Inadvertent removal of tubing prior to month 6 (Nervous system disorders) | 1 (1)
Inadvertent removal of tubing prior to month 6 (Social circumstances) | 1 (1)
Surgical removal of embedded accessory prior to month 6 (Surgical and medical procedures) | 1 (1)
Increased leakage due to migrating bumper (Product Issues) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT05288556/Prot_SAP_000.pdf